CLINICAL TRIAL: NCT00907036
Title: A Phase II Study of Reduced Intensity Sibling Allogeneic Transplantation for Relapsed, Chemosensitive, PET-positive Hodgkin Lymphoma
Brief Title: Fludarabine Phosphate, Melphalan, and Alemtuzumab Followed by Donor Stem Cell Transplant in Treating Patients With Relapsed Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CRUK-ReACH; CDR0000640500 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2008-004956-60; EU-20928; UCL/08/0122
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Alemtuzumab; Cyclosporine; fludarabine phosphate; Melphalan

INTERVENTIONS:
Biological: alemtuzumab
Biological: donor lymphocytes
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: melphalan
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. Also, monoclonal antibodies, such as alemtuzumab, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine before and after the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them (called graft-versus-tumor effect). Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

PURPOSE: This phase II trial is studying the side effects of fludarabine phosphate, melphalan, and alemtuzumab followed by donor stem cell transplant in treating patients with relapsed Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To document the toxicity, feasibility, and survival after reduced-intensity conditioning followed by allogeneic hematopoietic stem cell transplantation from a matched sibling donor in patients with relapsed, chemosensitive Hodgkin lymphoma.

OUTLINE: This is a multicenter study.

* Reduced-intensity conditioning: Patients receive fludarabine phosphate IV on days -7 to -3, melphalan IV over 30 minutes on day -2, and alemtuzumab IV on day -1.
* Transplantation: Patients undergo donor stem cell infusion on day 0.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV or orally on days -1 to 60, followed by a taper until 3 months post-transplantation, in the absence of GVHD.
* Donor-lymphocyte infusion (DLI): DLI is used for the eradication of mixed chimerism and for the management of residual or relapsed disease. If necessary, patients undergo DLI every 3 months until the desired endpoint is achieved or GVHD develops.

After completion of study therapy, patients are followed up every 3 months for 3 years.

This study is peer reviewed and funded or endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of Hodgkin lymphoma, meeting all of the following criteria:

  * Achieved partial or complete remission (using standard criteria) after salvage chemotherapy
  * Relapsed after first remission with residual fludeoxyglucose F 18-avid lesions
* Available HLA-matched sibling donor

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Creatinine clearance ≥ 50 mL/min (measured by EDTA clearance or 24-hour urine collection)
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* LVEF ≥ 40%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months (or 3 months for women) after completion of study therapy
* No other malignancy within the past 5 years except for nonmelanoma skin tumors or stage 0 (in situ) cervical carcinoma
* No HIV positivity
* No symptomatic respiratory compromise
* No concurrent serious medical condition that would preclude transplantation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior high-dose therapy or allograft

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2009-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival

SECONDARY OUTCOMES:
Donor engraftment rates, including chimerism at 3 and 6 months
Non-relapse mortality at 100 days and at 1 and 2 years post-transplant
Incidence of grade II-IV toxicity as assessed by NCI CTCAE v3.0
Incidence, severity, and timing of graft-vs-host disease
Response rates
Relapse rates
Response to donor lymphocyte infusions
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Karl Peggs, MD, Principal Investigator — University College London (UCL) Cancer Institute